CLINICAL TRIAL: NCT05419960
Title: Audio-vestibular Evaluation of Children and Young Adults With Osteogenesis Imperfecta
Acronym: AVOI
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220305; 2022-A00375-38 (Other: IDRCB Number)
Record Dates: First submitted 2022-05-12; First posted 2022-06-15 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis imperfecta; Vestibular deficits; Correlation between vestibular impairment and radiological findings; Bone abnormalities; Severity of the deafness
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients between the ages of 12-20 years with a diagnosis of Osteogenesis Imperfecta of any type and followed by a physician at the Centre de Référence des Maladies Rares des maladies osseuses constitutionnelles (CRMR OI) of Hôpital Necker-Enfants malades.
  Interventions: Diagnostic Test: Vestibular Assessment; Diagnostic Test: Petrous bone Computed Tomography (CT); Diagnostic Test: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Vestibular Assessment — During the usual hearing assessment (immittance testing and pure-tone and speech audiometry) carried out by patients, a vestibular assessment will be done for the study to detect vestibular disorders:
  * Videonystagmography (VNG) Is the study of eye movement with the help of infrared googles.
  * Subjective Visual Vertical (SVV) The patient is asked to orient a line on the vertical axis.
  * Video Head Impulse Test (vHIT)
  * Cervical and Ocular Vestibular Evoked Myogenic Potential (cVEMP and oVEMP)
Diagnostic Test: Petrous bone Computed Tomography (CT) — For patients diagnosed with hearing loss, whether conductive, mixed, and/or a vestibular deficit, a CT scan (without injection) will be proposed for their care.
  Petrous bone Computed Tomography (CT) is an imaging technique used as the standard method of evaluation of the boney structures in the ear.
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Patients that have done a CT and for who CT results was abnormal, will additionally require an MRI for their standard care.
  Magnetic Resonance Imaging (MRI) is an imaging technique used as the standard method of evaluation of the cochlear, retrocochlear and central and peripheral nervous system. An injection of Gadolinium contrast media will be used to enhance certain recordings.

SUMMARY:
The aim is to determine whether vestibular deficits are present in OI, then to establish whether a correlation exists between genetic type, severity of OI and audiovestibular phenotype. OI patients aged 12 to 20 years will undergo an audiometric, immittance, and vestibular assessment. When hearing loss is conductive or mixed or in cases where vestibular deficits are identified, a CT scan without injection will be performed. In case of sensorineural hearing loss or abnormal CT results, an MRI will be performed.

DETAILED DESCRIPTION:
Osteogenesis Imperfecta (OI), or Lobstein's disease, is a form of congenital osteoporosis, with a prevalence between 1/10,000 and 1/20,000 in France. As of 1979, four phenotypes have been described according to severity: moderate (type I), lethal (type II), severe (type III), and moderate-to-severe (type IV). OI exhibits phenotypic and genotypic variability, however, to date no correlations have been established between specific mutations and clinical presentation.

There is a well-established association between OI and hearing loss, however, the reported prevalence of hearing loss varies between 2% to 94.1%.

In patients with OI, Computed Tomography (CT) has revealed bone demineralization that progresses with age.

The extent of the hypodense areas on the CT corresponds to the type of hearing loss: conductive hearing loss is associated with lesions of the fissula ante fenestram and round and oval windows while mixed hearing loss is associated with additional retrofenestral lesions. Severity of hearing loss is positively correlated with OI-related bone damage in the petrous bone. Magnetic Resonance Imaging (MRI) has also revealed in the pericochlear lesions with soft tissue hypersignal and enhancement on contrast medium injection in the otic capsule. Bone demineralization has also been linked to vestibular deficits, and some studies have reported correlations between Osteogenesis Imperfecta and vestibular deficits in adult patients, however, this relationship is less clear.

The aim of the study is to determine whether vestibular deficits are also present in OI. Furthermore, the study will aim to establish whether a correlation exists between genetic type, severity of OI and audiovestibular phenotype. OI patients aged 12 to 20 years will be recruited and an audiometric, immittance, and vestibular assessment (videonystagmography, video Head Impulse Test (vHIT), vestibular evoked muscular potentials (cVEMP)) will be performed during their annual visit to the Centre de Référence des Maladies Rares des maladies osseuses constitutionnelles (henceforth CRMR OI) of Hôpital Necker-Enfants malades, Paris, France. When hearing loss is conductive, or mixed or in cases where vestibular deficits are identified, a CT scan without injection will be performed for the care. In case of sensorineural hearing loss, or abnormal CT results, an MRI will be proposed for the care. The investigation team will try to establish if there is a significant association between OI and vestibular deficit, and if so, whether the degree of vestibular impairment is correlated to radiological findings with respect to bone abnormalities, as well as the type and severity of the deafness.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 12-20 years at the time of inclusion
* Diagnosis of Osteogenesis Imperfecta of any type
* Currently followed by a physician at the CRMR OI
* Information and non-opposition of major patients, holders of parental authority and minor patients to participate in the study

Exclusion Criteria:

* Patients with hearing loss of alternate origin e.g. Cochlear nerve deficiency, atresia, etc.
* Neurological or developmental deficits limiting participation
* Cervico-occipital instability e.g. Chiari's malformation
* Limitations in mobility of the spine e.g. scoliosis, spinal fractural fusion
* Ophthalmologic pathologies e.g. strabism or severe refraction disorder
* Patients under AME (State Medical Aid)
* Protected adult patients, adults unable to express their consent, pregnant or breastfeeding women

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and young adults with a diagnosis of Osteogenesis Imperfecta of any type and followed by a physician at the Centre de Référence des Maladies Rares des maladies osseuses constitutionnelles (CRMR OI) of Hôpital Necker-Enfants malades.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2027-12-22 (Estimated); Study Completion 2027-12-22 (Estimated)

PRIMARY OUTCOMES:
Central Vestibular Function | 24 months
  Is evaluated by videonystagmography (VNG). The purpose of this test battery is to separate the vestibular disorders from disorders of the central neural system.
  Clinical norms will be applied to determine whether the exam is either within normal limits or abnormal.
  Research of eventual vestibular disorder to determine if vestibular disorders can be linked to Osteogenesis Imperfecta.
Subjective Visual Vertical (SVV) | 24 months
  Utricular Function Research of eventual vestibular disorder to determine if vestibular disorders can be linked to Osteogenesis Imperfecta.
  The patient is asked to orient a line on the vertical axis. An angle of 3 degrees from the vertical indicates an otolithic utricular disorder.
  Clinical norms will be applied to determine whether the exam is either within normal limits or abnormal.
Ocular Vestibular Evoked Myogenic Potential (oVEMP) | 24 months
  Utricular Function Research of eventual vestibular disorder to determine if vestibular disorders can be linked to Osteogenesis Imperfecta.
  The oVEMP assesses utricular function and reflects the function of the vestibular nuclei and the crossed vestibulo-ocular reflex (VOR) pathways, mostly contained in the medial longitudinal fasciculus (MLF).
  Clinical norms will be applied to determine whether the exam is either within normal limits or abnormal.
Semi-circular canal function | 24 months
  Video Head Impulse Test (vHIT). The vHIT assesses the vestibular ocular reflex linked to the semi-circular canal function when stimulated at a high frequency.
  Clinical norms will be applied to determine whether the exam is either within normal limits or abnormal.
  Research of eventual vestibular disorder to determine if vestibular disorders can be linked to Osteogenesis Imperfecta.
Cervical Vestibular Evoked Myogenic Potential (cVEMP) | 24 months
  Saccular Function Research of eventual vestibular disorder to determine if vestibular disorders can be linked to Osteogenesis Imperfecta.
  The cVEMP assesses the saccular function via the saccular cervical reflex (sternocleidomastoid muscle's activation secondary to saccular auditory stimulation).
  Clinical norms will be applied to determine whether the exam is either within normal limits or abnormal.
  The otolith organs are comprised of the vestibular saccule and utricule. The cVEMP assesses the saccular function via the saccular cervical reflex (sternocleidomastoid muscle's activation secondary to saccular auditory stimulation).
  Clinical norms will be applied to determine whether the exam is either within normal limits or abnormal.
  Research of eventual vestibular disorder to determine if vestibular disorders can be linked to Osteogenesis Imperfecta.

SECONDARY OUTCOMES:
Immittance testing | 24 months
  Audiological phenotype Immittance testing can indicate whether middle ear structures are in tact
  * Middle ear pressure and compliance of the tympanic membrane
  * Ipsilateral acoustic reflex thresholds
Pure-tone audiometry | 24 months
  Audiometry performance Pure tone audiometry is used to establish the type and degree of hearing loss. This measure is important to characterize the audiological phenotype. Hearing thresholds established in air and bone conduction between 250-8000Hz in each ear.
  Pure tone audiometry assessed as normal or abnormal Audiometry is considered abnormal if any threshold is greater than or equal to 25 dB HL.
Speech Audiometry | 24 months
  Audiometry performance Speech audiometry is used to establish the lowest intensity level in dB at which the patient can comprehend 50% of speech. This measure is important to confirm reliability of the pure tone audiometry, and to confirm that speech is both audible and intelligible.
  Speech audiometry assessed as normal or abnormal.
Severity of OI | 24 months
  OI medical diagnosis. The OI diagnosis is clinical, based on the following signs: ligament laxity, bluish discoloration of the sclera, hearing loss, vascular tissue abnormalities, hemostatic disorder, elevated basal metabolic rate, renal disorder, neurological disorder, history family.
  Depending on symptom severity, OI patient's diagnosis will be classified into on of four phenotypes : moderate (type I), lethal (type II), severe (type III), and moderate-to-severe (type IV).
Petrous bone Computed Tomography (CT) | 24 months
  CT is used to evaluate the presence and localization of petrous bone anomalies, for patients with conductive or mixed hearing loss and/or vestibular deficits.
Magnetic Resonance Imaging (MRI) | 24 months
  MRI is used to evaluate the presence and characteristics of anomalies of inner ear soft tissues, for patients with sensorineural hearing loss and for patients with abnormal CT scan results.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Loundon, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Marine Parodi, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No